CLINICAL TRIAL: NCT03257670
Title: Prospective Randomized Trial Comparing Treatment of Dyspareunia With Fractional CO2 Laser Therapy Versus 4% Topical Lidocaine Gel in the Setting of Breast Cancer Survivors.
Brief Title: Fractional CO2 Laser Therapy Versus 4% Topical Lidocaine Gel for Dyspareunia in Breast Cancer Survivors
Acronym: BCLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: Syneron Candela (Industry)
Responsible Party: Principal Investigator, James Whiteside, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC Laser
Record Dates: First submitted 2017-06-23; First posted 2017-08-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Dyspareunia
Keywords: Dyspareunia; Laser; CO2; Breast Cancer; Vaginal Atrophy; Lidocaine
MeSH Terms: conditions — Dyspareunia; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to two treatment cohorts (each with 35 patients): (1) treatment with the CO2RE laser or; (2) treatments of 4% aqueous lidocaine applied to the vulvar vestibule for 3 minutes before vaginal penetration. Both cohorts will have four follow-up assessments following initiation of treatment: (1) One-week post treatment initiation; (2) 1-month post treatment initiation; (3) 3-months post treatment initiation and; (4) 6-months post laser-only treatment initiation. At the 3-month assessment, subjects in the lidocaine arm will be allowed to try the CO2RE laser therapy. In doing this, an imbedded crossover trial is included that will allow assessment of subject decision-satisfaction between the two therapy approaches. The primary outcome will be the overall and lubrication, satisfaction, and pain domain scores on the Female Sexual Function Index instrument. Secondary outcomes will be other validated pain and pelvic floor symptom instruments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CO2RE Laser (Active Comparator): This group will undergo vaginal CO2 laser therapy for a total of three (3) treatments with one month between treatments.
  Interventions: Device: CO2RE fractional laser therapy
- 4% Topical Lidocaine Gel (Active Comparator): This group will be given 4% topical lidocaine gel to take home. The patient will apply the 4% lidocaine gel to the outside and opening of the vagina for 3 minutes before vaginal penetration. The patient will continue using the numbing gel prior to vaginal penetration for the extent of the study (3 months).
  Interventions: Drug: 4% Topical Lidocaine Gel

INTERVENTIONS:
Drug: 4% Topical Lidocaine Gel — This group will be given 4% topical lidocaine gel to take home. The patient will apply the 4% lidocaine gel to the outside and opening of the vagina for 3 minutes before vaginal penetration. The patient will continue using the numbing gel prior to vaginal penetration for the extent of the study (3 months).
  Arms: 4% Topical Lidocaine Gel
Device: CO2RE fractional laser therapy — This group will undergo vaginal CO2 laser therapy for a total of three (3) treatments with one month between treatments.
  Arms: CO2RE Laser

SUMMARY:
This trial seeks to determine if therapy with a CO2 laser to the vagina is more effective than lidocaine to the opening of the vagina before intercourse to reduce painful intercourse in women who are breast cancer survivors. This study will also be looking at whether or not the CO2 laser improves pelvic floor function, bowel and bladder function, and sexual function before and after treatment.

DETAILED DESCRIPTION:
This is a randomized trial to determine the comparative effectiveness of the CO2RE laser device relative to topical lidocaine in treating dyspareunia among breast cancer survivors. The large and growing population of breast cancer survivors experience a significant burden of urogenital symptoms including dyspareunia. Several studies have evaluated the feasibility and effectiveness of CO2 lasers for the treatment of symptomatic vulvovaginal atrophy in postmenopausal women suggesting improvements in atrophy symptoms with favorable histological and microscopic changes. There is little know about the effectiveness of CO2 laser therapy in breast cancer survivors.

Patients who are breast cancer survivors experiencing dyspareunia and desiring intervention will be randomized to two cohorts: (1) Treatment with the CO2RE laser or (2) application of 4% aqueous lidocaine applied to the vulvar vestibule for 3 minutes before vaginal penetration. The primary outcome will be the overall as well as lubrication, satisfaction, and pain domain scores on the Female Sexual Function Index instrument. Secondary outcomes will be according to other validated pain and pelvic floor symptom instruments.

Following initiation of treatment, both groups will follow up at one-week, 1-month, 3-months, and 6-months. At the 3-month assessment, subjects in the lidocaine arm will be given the option to undergo CO2RE laser therapy. A combination of validated and non-validated physical exam and survey instruments will be utilized at each visit in order to assess pelvic floor function, bowel and bladder function, and sexual function before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included must be female breast cancer survivors over the age of 18, sexually active (at least 4 episodes of sexual intercourse per month), and find intercourse painful. Subjects must also be English speaking and able to give informed consent.

Exclusion Criteria:

* Subjects will be excluded if pregnant, has not had breast cancer, does not have painful intercourse secondary to treatment received for their breast cancer, is not English speaking, or lacks the ability to sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects must be female who have undergone treatment for breast cancer that have dyspareunia secondary to the treatment they received for breast cancer.
Enrollment: 70 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) score before and after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The Female Sexual Function Index (FSFI) is a survey instrument used to determine the level of sexual function or dysfunction in females. It is comprised of a 19 item questionnaire focused on sexual functioning. There are six domains assessed: desire, arousal, lubrication, orgasm, satisfaction, and pain. The subject is to consider each of the questions in the context of the previous 4 weeks. The scores of each of the domains are then calculated into a final score.
  Initial and follow-up assessments will allow comparisons across this instrument as well as all the secondary and other pre-specified outcome measures.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) score before and after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The Numeric Pain Rating Scale (NPRS) is a measure of pain intensity in adults.The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. Similar to the VAS, the NPRS is anchored by terms describing pain severity extremes. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").The NPRS can be administered verbally (therefore also by telephone) or graphically for self-completion. Scores range from 0-10 with higher numbers representing higher pain intensity.
Incontinence Severity Index (ISI) score before and after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The Incontinence Severity Index (ISI) consists of two questions, regarding frequency and amount of leakage. It categorizes urinary incontinence (UI) into none, slight, moderate, severe, and very severe. It assess the frequency (from 0-4): (0-never, 1-less than once a month, 2-a few times a month, 3-a few times a week, 4-every day and/or night ), and amount (from 0-3) of urine leakage: 0-none, 1-drops, 2-small splashes, 3-more. The index value is from 0-12 obtained by multiplying the numbers responded in the two questions with categories of urinary incontinence severity of: None (0), Slight (1-2), Moderate (3-6), Severe (8-9), Very severe (12).
3 Incontinence Questions (3-IQ) score before and after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The 3 Incontinence Questions (3-IQ) is a survey instrument that is used to determine if a patient has stress urinary incontinence (SUI), urge urinary incontinence (UUI), or mixed urinary incontinence (MUI). The subject is to consider each of the questions in the context of the previous 3 months.The first question asks if the patient has every leaked urine. The second question asks the patient to indicate if she has leaked urine with any of the following: activity, urge, or without activity or urge. The Third question asks which form of urinary leakage was most common. The response to question 3 is then used to determine if the patient has: 1) Stress only or mostly stress, 2) urge only or mostly urge, 3) other cause, or 4) mixed.
Colon Rectal Anal Distress Inventory (CRADI) score before and after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The Colon Rectal Anal Distress Inventory (CRADI) is a survey instrument used to determine the level and severity of bowel symptoms. It consists of 17 questions inquiring to specific questions regarding bowel symptoms. Total score out of 400, with higher scores indicating more bowel symptoms.
Patient Global Impression of Severity (PGI-S) score before treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The PGI-S are 1 question assessments of overall condition severity before implementation of therapy measured on a 7-point response scale.
Patient Global Impression of Improvement (PGI-I) score after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The Patient Global Impression of Improvement (PGI-I) is 1 question assessment of overall condition improvement since implementation of therapy measured on a 7-point response scale.
Satisfaction with Decision (SDS) score before and after treatment with topical lidocaine ointment or transvaginal CO2 laser among breast cancer survivors with dyspareunia. | 9 months
  The Satisfaction with Decision (SDS) was developed to measure patient satisfaction with health care decisions. The SDS is a 6-item questionnaire with a 5-point response scale with higher scores indicating higher overall satisfaction.

OTHER OUTCOMES:
Symptom inventory (number of voids/day, pads/day, etc.) | 9 months
  Symptom inventory (number of voids/day, pads/day, etc.) will be collected and available for comparison by cohort prior to and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James L Whiteside, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] Maiorino MI, Chiodini P, Bellastella G, Giugliano D, Esposito K. Sexual dysfunction in women with cancer: a systematic review with meta-analysis of studies using the Female Sexual Function Index. Endocrine. 2016 Nov;54(2):329-341. doi: 10.1007/s12020-015-0812-6. Epub 2015 Dec 7. PMID 26643312
- [Background] Mazzarello S, Hutton B, Ibrahim MFK, Jacobs C, Shorr R, Smith S, Ng T, Clemons M. Management of urogenital atrophy in breast cancer patients: a systematic review of available evidence from randomized trials. Breast Cancer Res Treat. 2015 Jul;152(1):1-8. doi: 10.1007/s10549-015-3434-z. Epub 2015 May 24. PMID 26003182
- [Background] Falk SJ, Bober S. Vaginal Health During Breast Cancer Treatment. Curr Oncol Rep. 2016 May;18(5):32. doi: 10.1007/s11912-016-0517-x. PMID 27074843
- [Background] Baumgart J, Nilsson K, Stavreus-Evers A, Kask K, Villman K, Lindman H, Kallak T, Sundstrom-Poromaa I. Urogenital disorders in women with adjuvant endocrine therapy after early breast cancer. Am J Obstet Gynecol. 2011 Jan;204(1):26.e1-7. doi: 10.1016/j.ajog.2010.08.035. Epub 2010 Oct 14. PMID 20950790
- [Background] Sinha A, Ewies AA. Non-hormonal topical treatment of vulvovaginal atrophy: an up-to-date overview. Climacteric. 2013 Jun;16(3):305-12. doi: 10.3109/13697137.2012.756466. Epub 2013 Jan 8. PMID 23215675
- [Background] Perino A, Calligaro A, Forlani F, Tiberio C, Cucinella G, Svelato A, Saitta S, Calagna G. Vulvo-vaginal atrophy: a new treatment modality using thermo-ablative fractional CO2 laser. Maturitas. 2015 Mar;80(3):296-301. doi: 10.1016/j.maturitas.2014.12.006. Epub 2014 Dec 25. PMID 25596815
- [Background] Salvatore S, Nappi RE, Zerbinati N, Calligaro A, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. A 12-week treatment with fractional CO2 laser for vulvovaginal atrophy: a pilot study. Climacteric. 2014 Aug;17(4):363-9. doi: 10.3109/13697137.2014.899347. Epub 2014 Jun 5. PMID 24605832
- [Background] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Background] Zerbinati N, Serati M, Origoni M, Candiani M, Iannitti T, Salvatore S, Marotta F, Calligaro A. Microscopic and ultrastructural modifications of postmenopausal atrophic vaginal mucosa after fractional carbon dioxide laser treatment. Lasers Med Sci. 2015 Jan;30(1):429-36. doi: 10.1007/s10103-014-1677-2. Epub 2014 Nov 20. PMID 25410301
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] Sandvik H, Hunskaar S, Seim A, Hermstad R, Vanvik A, Bratt H. Validation of a severity index in female urinary incontinence and its implementation in an epidemiological survey. J Epidemiol Community Health. 1993 Dec;47(6):497-9. doi: 10.1136/jech.47.6.497. PMID 8120507
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Background] Sung VW, Kauffman N, Raker CA, Myers DL, Clark MA. Validation of decision-making outcomes for female pelvic floor disorders. Am J Obstet Gynecol. 2008 May;198(5):575.e1-6. doi: 10.1016/j.ajog.2007.12.035. Epub 2008 Mar 7. PMID 18313632
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Sandvik H, Espuna M, Hunskaar S. Validity of the incontinence severity index: comparison with pad-weighing tests. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Sep;17(5):520-4. doi: 10.1007/s00192-005-0060-z. Epub 2006 Mar 18. PMID 16547687
- [Background] Brown JS, Bradley CS, Subak LL, Richter HE, Kraus SR, Brubaker L, Lin F, Vittinghoff E, Grady D; Diagnostic Aspects of Incontinence Study (DAISy) Research Group. The sensitivity and specificity of a simple test to distinguish between urge and stress urinary incontinence. Ann Intern Med. 2006 May 16;144(10):715-23. doi: 10.7326/0003-4819-144-10-200605160-00005. PMID 16702587